CLINICAL TRIAL: NCT04753827
Title: "L-Sandwich" Strategy in the True Coronary Bifurcation Lesions
Acronym: L-Sandwich
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HenanICE202102
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Intervention Model Description: Three different strategies for true bifurcation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group Stent only (Experimental): Stents were implanted in MV and SB respectively, and DKcrush or Culotte technology was selected according to the lesion characteristics.
  Interventions: Other: Drug eluting stent
- Experimental Group Stent+DCB (Experimental): The MV was stented and the SB were treated with just drug-coated balloon(DCB)
  Interventions: Other: Drug eluting stent; Other: Durg coated balloon
- Experimental Group L-Sandwich (Experimental): Stents were implanted in the MV and the shaft of side branch SB respectively, then a DCB was applied to the ostium of the SB
  Interventions: Other: Drug eluting stent; Other: Durg coated balloon

INTERVENTIONS:
Other: Drug eluting stent — Put a Drug eluting stent in the blood vessel
Other: Durg coated balloon — Put a Durg coated balloon in the blood vessel
  Arms: Experimental Group L-Sandwich; Experimental Group Stent+DCB

SUMMARY:
The treatment of coronary bifurcation lesions continue to remain challenges. Due to the complexity of the anatomical structure and the limitations of imaging, there are poor attachment and under-expansion of the stent at the branch ostium, which causes in-stent thrombosis and restenosis. The delayed re-endothelialization arise from multi-layer stents. The one-stent strategy causes the displacement of the plaques and ridges of the branch ostium, and thus insufficient blood flow to the branches. The "L-sandwich" strategy, stents were implanted in the main vessel(MV) and the shaft of side branch(SB) respectively, then a drug-coated balloon(DCB) was applied to the ostium of the SB, to improve the tedious operation process in true bifurcation lesions and reduce postoperative complications. The purpose of this study was to explore the feasibility, safety, and efficacy of the "sandwich" strategy.

DETAILED DESCRIPTION:
This is a study to evaluate the application of L-Sandwich in true bifurcation coronary artery disease.All eligible patients were randomly divided into three groups: experimental group 1: dual stent group: both main vessel(MV) and side branch(SB) were stented, and DK-Crush or Culotte were performed according to different pathological characteristics. Experimental group 2: single stent + drug-coated balloon（DCB）: stent was implanted in the MV, and only drug balloon was used in the SB.Experimental group 3: L-Sandwich : stent was implanted in the MV, and the branch was implanted 3-5mm away from the ostium，and the DCB was implanted in the ostium of the branch.IVUS+ angiography was used to guide the operation and evaluate the outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with true bifurcation disease with SB lesion length>25mm

Exclusion Criteria:

* SB diameter<2.5mm
* presence of cardiogenic shock or cardiopulmonary resuscitation
* Expected survival <1 year
* Allergy to indexed medications
* Intolerable to dual antiplatelet therapy
* pregnant
* Severe calcification needing rotational atherectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-10-03 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
main vessel late lumen loss | 6 months
  main vessel late lumen loss
Side branch late lumen loss | 6 months
  Side branch late lumen loss

SECONDARY OUTCOMES:
Target lesion failure rate | 30days
  Cardiac death,Target vessel MI,Target lesion revascularization
Target lesion failure rate | 6 months
  Cardiac death,Target vessel MI,Target lesion revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Muwei Li, MD, Study Chair — FF
Locations (1):
- Fuwai central China cardiovascular Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No
Others can obtain the individual participant data from the researcher by reasonable request